CLINICAL TRIAL: NCT06901154
Title: Influence of the 3D-sonographic Representation of the Fetal Face on the Health-conscious Behavior of Pregnant Women
Acronym: IN3D
Status: Not yet recruiting | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Marcus Riemer, MD, deputy director, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKGEB004
Record Dates: First submitted 2025-03-11; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pregnant women: pregnant women undergoing ultrasound

SUMMARY:
Studies have shown that ultrasound examinations during pregnancy have a short-term anxiety and stress-reducing effect, without having any influence on the mother-child bond or health-conscious behavior.

It has not yet been investigated to what extent the representation of the child's face alone achieves a lasting positive effect if the representation in 3D form were permanently available.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women undergoing ultrasound

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Influence on the health-conscious behavior | through study completion, an average of 3 months
  Measuring influence through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Riemer, MD, Principal Investigator — University Hospital of Halle

IPD SHARING:
Plan to Share IPD: Undecided